CLINICAL TRIAL: NCT06706531
Title: Additional Effects of Dry Needling With Conventional Physical Therapy Versus Conventional Physical Therapy in Plantar Fasciitis: a Randomized Control Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/53
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Plantar Fascitis
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment + Sham Dry needling (Active Comparator): Participants will receive standard treatment of plantar facitis along with sham dry needling
  Interventions: Procedure: Standard treatment; Procedure: Sham Dry needling
- Standard treatment + Dry needling (Experimental): Participants will receive standard treatment of plantar facitis along with dry needling
  Interventions: Procedure: Standard treatment; Procedure: Dry needling

INTERVENTIONS:
Procedure: Standard treatment — All participants received up to six treatment sessions at a frequency of twice per week over a 3-week period i.e. ultrasound (0.5 W/cm² of 3 MHz for 5 minutes over plantar aspect of foot), stretching exercises and strengthening exercises. The exercise pro
Procedure: Sham Dry needling — The sham dry needling group will also receive 6 sessions of sham dry needling on soleus, quadratus plantae, flexor digitorum brevis, and abductor halluces muscles for 5 minutes.Sterilized disposable stainless steel acupuncture needles of 0.25mm x 30mm will be used with depth of 20-55mm.The plantar and medial surface of the foot and ankle will be cleaned with alcohol. The sham dry needling will be performed for 5 minutes.
  Arms: Standard treatment + Sham Dry needling
Procedure: Dry needling — The dry needling group will receive 6 sessions of dry needling using a standardized trigger point protocol on soleus, quadratus plantae, flexor digitorum brevis, and abductor halluces muscles for 5 minutes. Sterilized disposable stainless steel acupuncture needles of 0.25mm x 30mm will be used with depth of 20-55mm. The calf, plantar and medial surface of the foot and ankle will be cleaned with alcohol. Following insertion, needles will be manipulated bi-directionally to elicit a sensation of aching, tingling, deep pressure, heaviness or warmth. The needles will then left in situ for 5 minutes.
  Arms: Standard treatment + Dry needling

SUMMARY:
This study is a randomized controlled trial and the purpose of this study is to determine the effects of dry needling with conventional physical therapy versus conventional physical therapy on gait parameters in plantar fasciitis: a randomized control trial.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of dry needling with conventional physical therapy versus conventional physical therapy on gait parameters in plantar fasciitis Outcomes variables of Pain , Ankle ROM, gait parameters and activities of daily living in adults (age : 40-60 years ) will be determined using:

1. Numeric pain rating scale
2. Goniometer
3. 30 meter walk test
4. foot and ankle ability measure FAAM Data will be before and after the intervention protocol for each participant. Data collection procedure: Participants of interest would be approached and explained about the research. Informed written consent will be taken. Pre and post intervention scores will be recorded.

ELIGIBILITY:
Inclusion criteria:

* Age 40-60 years
* Both genders
* Plantar heel pain for longer than 3 months
* Pain score at least or less than 8 on the numeric pain (NPRS)
* Clinical diagnosis of unilateral PF in accordance with the clinical practice guidelines from the Orthopaedic Section of the American Physical Therapy Association APTA:
* Plantar medial heel pain: most noticeable with initial steps after a period of inactivity but also worse following prolonged weight bearing
* Heel pain precipitated by a recent increase in weight bearing activity
* Pain with palpation of the proximal insertion of the plantar fascia
* Positive windlass test
* Negative tarsal tunnel tests
* Limited active and passive talocrural joint dorsiflexion range of motion
* Abnormal foot posture index score
* High body mass index in nonathletic individuals

Exclusion criteria:

* Positive ankle drawer tests
* Pregnant womwn, mental illness, immune suppressed patients, thrombocytopenia, anti-coagulant therapy patients and post-mastectomy
* Congenital abnormalities of foot
* A history of surgery to the ankle, foot or lower leg
* Other causes of heel pain (including tarsal tunnel syndrome, calcaneal fracture, ankle or foot instability, arthritis of the foot or ankle, rheumatoid arthritis, spondyloarthropathy, gout,peripheral neuropathy )
* Presented with 2 or more positive neurologic signs consistent with nerve root compression

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 3 weeks
  Pain will be measured on Numerical Pain rating scale. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
The Foot and Ankle Ability Measure (FAAM) | 3 weeks
  It is a self-report outcome instrument developed to assess physical function for individuals with foot and ankle related impairments .The response to each item on the ADL subscale is scored from 4 to 0, with 4 being 'no difficulty' and 0 being 'unable to do'
Gait speed: | 3 weeks
  Gait speed = Distance (m) / time (s)
Cadence | 3 weeks
  Cadence (steps/min) = steps counted x 60 / time (s)
Cycle length | 3 weeks
  Cycle time (s) = time (s) x 2/steps counted
Stride length | 3 weeks
  SL (m) = speed (m/s) x cycle time (s)
Range of motion | 3 weeks
  Ankle range will be measured with goniometer

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan